CLINICAL TRIAL: NCT01159795
Title: Investigating Type I and Type III Interferon Responses in Infants With Respiratory Syncytial Virus
Brief Title: Studying Innate Immune Responses in Infants With Bronchiolitis
Status: Terminated | Type: Observational
Why Stopped: Awaiting further funding
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 10/H0707/24
Record Dates: First submitted 2010-07-06; First posted 2010-07-09 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2012-04

CONDITIONS: Bronchiolitis
Keywords: Respiratory Syncytial Virus; Infant; Interferon
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma - cytokines Blood EDTA - DNA Blood PAXgene tube - RNA Nasal lining fluid - cytokines Nasal mucosal lining - RNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to establish whether impaired innate immune responses are associated with severity of Respiratory syncytial virus (RSV) infection.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) causes a spectrum of illness in healthy infants, ranging from asymptomatic infection to life threatening bronchiolitis with respiratory failure. The reasons for the differences in clinical presentation remain unknown. Interferons are natural antiviral factors and components of the innate immune response, which play a role in limiting viral replication.

We postulate that differences in clinical severity of RSV infection may be due to innate immune differences in the production of type I and III interferons (innate interferons). To test this hypothesis, we will recruit infants with mild, moderate and severe RSV bronchiolitis and compare production of innate interferons in blood and respiratory samples, using quantitative and functional analysis. We will determine whether interferon responses differ across a spectrum of clinical severity, and will relate them to viral load.

To establish whether defects in interferon production persist in those infants with severe infection, we will retest them following recovery and measure interferon responses after challenge with live RSV. Demonstrating a persisting defect may suggest a genetically determined defect requiring further investigation. Identification of the mechanisms of severe disease in patients without known risk-factors could lead to targeted therapy to prevent or treat severe disease.

ELIGIBILITY:
Inclusion Criteria:

* Bronchiolitis
* Infant

Exclusion Criteria:

* Age over 1 year
* Underlying chronic lung disease, prematurity, congenital heart disease

Ages: 6 Weeks to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants presenting with bronchiolitis presenting to St Mary's Hospital, London
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Nasal and blood interferon alpha, beta, lambda levels(protein level and gene expression) | At presentation (average = day 4 of symptoms)
  Interferon alpha, beta and lambda protein levels will be measured by ELISA and gene expression by quantitative real-time PCR, on paired nasal and blood samples.

SECONDARY OUTCOMES:
RSV viral load | At presentation (average = day 4 of symptoms)
  RSV viral load will be measured by quantitataive real-time PCR on nasal epithelium samples.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levin, FMed Sci, Principal Investigator — Department of Paediatrics, Imperial College London
Locations (1):
- St Mary's Hospital, London, United Kingdom